CLINICAL TRIAL: NCT03935152
Title: Oral Dydrogesterone as Adjunctive Therapy in the Management of Preterm Labor: A Randomized, Double Blinded, Placebo-controlled Trial
Brief Title: Oral Dydrogesterone in the Management of Preterm Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 286/2019
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dydrogesterone (Active Comparator): dydrogesterone 10 mg by mouth every 8 hours until delivery
  Interventions: Drug: Dydrogesterone
- Placebo (Placebo Comparator): placebo by mouth every 8 hours until delivery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dydrogesterone — dydrogesterone capsule
  Arms: Dydrogesterone
Drug: placebo — placebo capsule
  Arms: Placebo

SUMMARY:
This study evaluates the addition of oral dydrogesterone to standard treatment in the treatment of preterm labor. Half of participants will receive oral dydrogesterone and standard treatment, while the other half will receive oral placebo and standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy with gestational age 24-33 weeks 6 days
* preterm labor
* received treatment with tocolysis and corticosteroids

Exclusion Criteria:

* conditions that need immediate delivery such as fetal distress, chorioamnionitis
* have medical complications such as heart disease, seizure
* fetal anomalies
* cervical dilatation more than 5 cm
* allergy to dydrogesterone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 48 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
latency period | 13 weeks
  time from preterm labor to delivery

SECONDARY OUTCOMES:
preterm delivery less than 34 weeks | 10 weeks
  percentage of delivery less than 34 weeks
preterm delivery less than 37 weeks | 13 weeks
  percentage of delivery less than 37 weeks
neonatal complications | 13 weeks
  percentage of newborn with RDS, IVH, NEC, death
side effects | 13 weeks
  percentage of side effects such as headache, nausea/vomiting
compliance | 13 weeks
  percentage of complete drug use
satisfaction | 13 weeks
  percentage of good satisfaction
Time to the recurrence of uterine contractions | 13 weeks
  Time to the recurrence of uterine contractions

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University, Faculty of Medicine, Department of Obstetrics and Gynecology
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 171: Management of Preterm Labor. Obstet Gynecol. 2016 Oct;128(4):e155-64. doi: 10.1097/AOG.0000000000001711. PMID 27661654
- [Background] Blencowe H, Cousens S, Chou D, Oestergaard M, Say L, Moller AB, Kinney M, Lawn J; Born Too Soon Preterm Birth Action Group. Born too soon: the global epidemiology of 15 million preterm births. Reprod Health. 2013;10 Suppl 1(Suppl 1):S2. doi: 10.1186/1742-4755-10-S1-S2. Epub 2013 Nov 15. PMID 24625129
- [Background] Norwitz ER, Caughey AB. Progesterone supplementation and the prevention of preterm birth. Rev Obstet Gynecol. 2011 Summer;4(2):60-72. PMID 22102929
- [Background] Yasuda K, Sumi GI, Murata H, Kida N, Kido T, Okada H. The steroid hormone dydrogesterone inhibits myometrial contraction independently of the progesterone/progesterone receptor pathway. Life Sci. 2018 Aug 15;207:508-515. doi: 10.1016/j.lfs.2018.07.004. Epub 2018 Jul 4. PMID 29981319
- [Background] Schindler AE, Campagnoli C, Druckmann R, Huber J, Pasqualini JR, Schweppe KW, Thijssen JH. Classification and pharmacology of progestins. Maturitas. 2008 Sep-Oct;61(1-2):171-80. doi: 10.1016/j.maturitas.2008.11.013. PMID 19434889
- [Result] Borna S, Sahabi N. Progesterone for maintenance tocolytic therapy after threatened preterm labour: a randomised controlled trial. Aust N Z J Obstet Gynaecol. 2008 Feb;48(1):58-63. doi: 10.1111/j.1479-828X.2007.00803.x. PMID 18275573
- [Result] Arikan I, Barut A, Harma M, Harma IM. Effect of progesterone as a tocolytic and in maintenance therapy during preterm labor. Gynecol Obstet Invest. 2011;72(4):269-73. doi: 10.1159/000328719. Epub 2011 Nov 12. PMID 22086108
- [Result] Choudhary M, Suneja A, Vaid NB, Guleria K, Faridi MM. Maintenance tocolysis with oral micronized progesterone for prevention of preterm birth after arrested preterm labor. Int J Gynaecol Obstet. 2014 Jul;126(1):60-3. doi: 10.1016/j.ijgo.2014.01.019. Epub 2014 Apr 3. PMID 24807871
- [Result] Areeruk W, Phupong V. A randomized, double blinded, placebo controlled trial of oral dydrogesterone supplementation in the management of preterm labor. Sci Rep. 2016 Feb 9;6:20638. doi: 10.1038/srep20638. PMID 26856618
- [Derived] Thongchan S, Phupong V. Oral dydrogesterone as an adjunctive therapy in the management of preterm labor: a randomized, double blinded, placebo-controlled trial. BMC Pregnancy Childbirth. 2021 Jan 28;21(1):90. doi: 10.1186/s12884-021-03562-6. PMID 33509129